CLINICAL TRIAL: NCT04046289
Title: Effects of 6-Month Probiotics and Calcium Supplementation During Childhood on Growth, Development, and Metabolic Parameters in Adolescents: A 10-Year Follow-up Study
Brief Title: Effects of Probiotics and Calcium Supplementation on Growth, Development, and Metabolic Parameters
Acronym: PROBIOCAL
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Collaborators: SEAMEO Regional Centre for Food and Nutrition (Other); Wageningen University (Other)
Responsible Party: Principal Investigator, Rina Agustina, Principal Investigator, Indonesia University
Other Study IDs: probiocal
Record Dates: First submitted 2019-08-01; First posted 2019-08-06 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Stunting; Obesity; Cognitive Function 1, Social; Depression; Behavior; Dyslipidemias; Insulin Resistance; Permeability; Increased
MeSH Terms: conditions — Growth Disorders; Obesity; Depression; Behavior; Dyslipidemias; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Low Calcium: low calcium milk of 180 ml, twice daily for 24 weeks
  Interventions: Dietary Supplement: Low Calcium Milk
- Regular Calcium: regular calcium milk of 180 ml, twice daily for 24 weeks
  Interventions: Dietary Supplement: Regular Calcium Milk
- Probiotic 1: regular calcium milk of 180 ml + probiotic, twice daily for 24 weeks
  Interventions: Dietary Supplement: Probiotic 1
- Probiotic 2: regular calcium milk of 180 ml + probiotic, twice daily for 24 weeks
  Interventions: Dietary Supplement: Probiotic 2

INTERVENTIONS:
Dietary Supplement: Low Calcium Milk — 50 mg calcium/day
  Groups: Low Calcium
Dietary Supplement: Regular Calcium Milk — 400 mg/day
  Groups: Regular Calcium
Dietary Supplement: Probiotic 1 — regular calcium milk + probiotic
  Groups: Probiotic 1
Dietary Supplement: Probiotic 2 — regular calcium milk + probiotic
  Groups: Probiotic 2

SUMMARY:
Stunting is still a major problem in developing countries, including Indonesia, and has been associated with impaired development. Stunted children have also a higher risk of metabolic syndrome in adulthood. The gut microbiota, as a part of intestinal integrity, may promote intake of nutrient during childhood. Probiotics supplementation may optimize the balance of gut microbiota and further improve child growth during the window period. Furthermore, calcium could also improve child growth by increasing the resistance to intestinal infection. However, the long-term effects of gut microbiota optimization during childhood using probiotics and calcium on growth, development, and the metabolic condition has not widely studied.

DETAILED DESCRIPTION:
This study was a 10-year follow-up study of randomized controlled trials of 6-month probiotics and calcium supplementation of Lactobacillus reuteri DSM 17938 or Lactobacillus casei CRL 431 in children aged 1-6 years (n=494) living in urban low socioeconomic communities of East Jakarta in 2007-2008. We re-enrolled the subjects to assess the long-term effects of probiotics and calcium supplementation on growth, development, and metabolic parameters at the age of 11-17 years.

Healthy children (n = 238) were included in this follow-up study. Each subject previously assigned to one intervention group: low-lactose milk with a low calcium content (LC = 53), a regular calcium content (RC = 70), regular calcium with L. reuteri DSM 17938 (n = 55), and regular calcium with L. casei CRL 431 (n = 60).

Anthropometric measurements were performed by measuring the weight and height of the subjects, and further combining the results to report BMI-for-age z-score. Height was also plotted to the chart of the World Health Organization (WHO) Child Growth Standards. Gut integrity was assessed with the lactulose-mannitol ratio using high-performance liquid chromatography (HPLC) method. Cognitive function, symptoms related to depression, behaviour, and serum brain-derived neurotrophic factors (BDNF) of the adolescents were evaluated used to investigate the effects of supplementation on development. We quantified lipid profile and Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) as metabolic parameters using the vein blood sample. The metabolic parameters were measured in at least three groups of intervention.

ELIGIBILITY:
Inclusion Criteria at the previous clinical trial:

* Apparently healthy children aged 1-6 years, with emphasize on aged 2-5 years, living permanently in low socio-economic urban areas of East Jakarta for at least six months
* Parents are willing to sign the informed consent and give the supplements to the children for six months
* Capable and willing to drink liquid milk with a straw (acceptance to be tested at the screening by providing a sample drink and placebo straw to be consumed under supervision for two days)

Exclusion Criteria at the previous clinical trial:

* Calcium intake exceeding 75% of the Recommended Dietary Allowance (RDA) for calcium (<375 mg/d) based on a Food Frequency Questionnaire
* Currently breastfed children
* Siblings of already included children that are living in the same household, except if it is a twin sibling
* Severely malnourished with or without edema (weight-for-height Z-score of <-3.00 SD)
* Symptoms of chronic/congenital diseases and disabilities, suspected Tuberculosis by clinical examination, and/or history of allergic disease.
* Taking (any) antibiotics during 2 weeks prior to the start of the study (children will be included after 3 weeks of last antibiotic intake
* Participation in another clinical trial at the same time or 2 months prior to the start of this study
* Both mothers and other caregivers present in the family are illiterate

Inclusion criteria of follow-up study:

* Healthy adolescent participated in the previous trial study willing to take part in the follow-up study

Exclusion criteria of follow-up study:

* History of type 1 diabetes
* Taking the cholesterol-lowering drug, an anti-diabetic drug, or oral corticosteroid for more than 2 consecutive weeks in the last 3 months
* Pregnant

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Low-socioeconomic urban communities representing flooding and non-flooding areas of East Jakarta, Indonesia.
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2019-01-26 (Actual); Primary Completion 2019-03-03 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Child's linear growth the age of 11-17 years | January - March 2019
  Height-for-age z-score based on the WHO Child Growth Standards.
Child's height at the age of 11-17 years | January - March 2019
  Height in meters.
Child's weight at the age of 11-17 years | January - March 2019
  Weight in kilograms.
Child's nutritional status at the age of 11-17 years | January - March 2019
  BMI-for-age z-score based on the WHO Child Growth Standards. BMI was calculated from height and weight measurement.

SECONDARY OUTCOMES:
Gut integrity at the age of 11-17 years | January - March 2019
  Lactulose-mannitol ratio was calculated by dividing percent excretion of lactulose with percent excretion of mannitol.
Cognitive function assessed using Raven's Progressive Matrices at the age of 11-17 years | January - March 2019
  Raven's Progressive Matrices (RPM) was administered by psychologists. Raw score of RPM was used to evaluate adolescents' cognition.
Symptoms related to depression assessed using Children Depression Inventory at the age of 11-17 years | January - March 2019
  Children Depression Inventory (CDI) was a self-assigned questionnaire and the total score of CDI with a range between 0 - 54 (lower, better) was used to evaluate the symptoms related to depression among adolescents.
Behaviour assessed using Strength and Difficulties Questionnaire at the age of 11-17 years | January - March 2019
  Strength and Difficulties Questionnaire (SDQ) was a self-assigned questionnaire and the total difficulties score of SDQ with a range between 0 - 50 (lower, better) was used to evaluate the behaviour among adolescents.
Serum BDNF at the age of 11-17 years | January - March 2019
  Serum BDNF in pg/ml was quantified using ELISA method
Triglyceride level at the age of 11-17 years | January - March 2019
  Triglyceride level in milligrams per decilitre.
High-density lipoprotein level at the age of 11-17 years | January - March 2019
  High-density lipoprotein level in milligrams per decilitre.
Low-density lipoprotein level at the age of 11-17 years | January - March 2019
  Low-density lipoprotein level in milligrams per decilitre.
Fasting insulin level at the age of 11-17 years | January - March 2019
  Fasting insulin level in μU per millilitre
Fasting glucose level at the age of 11-17 years | January - March 2019
  Fasting glucose level in milligrams per decilitre.
HOMA-IR at the age of 11-17 years | January - March 2019
  HOMA-IR was quantified by multiplying fasting insulin level with fasting glucose level.

CONTACTS AND LOCATIONS:
Overall Officials: Rina Agustina, PhD, Principal Investigator — HNRC IMERI; Department of Nutrition, Faculty of Medicine, Universitas Indonesia
Locations (1):
- Human Nutrition Research Center, Indonesian Medical Education Research Institute; and Department of Nutrition, Faculty of Medicine, Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Agustina R, Kok FJ, van de Rest O, Fahmida U, Firmansyah A, Lukito W, Feskens EJ, van den Heuvel EG, Albers R, Bovee-Oudenhoven IM. Randomized trial of probiotics and calcium on diarrhea and respiratory tract infections in Indonesian children. Pediatrics. 2012 May;129(5):e1155-64. doi: 10.1542/peds.2011-1379. Epub 2012 Apr 9. PMID 22492764
- [Background] Agustina R, Bovee-Oudenhoven IM, Lukito W, Fahmida U, van de Rest O, Zimmermann MB, Firmansyah A, Wulanti R, Albers R, van den Heuvel EG, Kok FJ. Probiotics Lactobacillus reuteri DSM 17938 and Lactobacillus casei CRL 431 modestly increase growth, but not iron and zinc status, among Indonesian children aged 1-6 years. J Nutr. 2013 Jul;143(7):1184-93. doi: 10.3945/jn.112.166397. Epub 2013 May 22. PMID 23700339
- [Derived] Agustina R, Rianda D, Setiawan EA. Relationships of Child-, Parents-, and Environment-Associated Determinants with Diet Quality, Physical Activity, and Smoking Habits Among Indonesian Urban Adolescents. Food Nutr Bull. 2022 Mar;43(1):44-55. doi: 10.1177/03795721211046145. Epub 2021 Oct 21. PMID 34670443
- [Derived] Setiawan EA, Rianda D, Kadim M, Meilianawati, Susanto F, Kok FJ, Shankar AH, Agustina R. Tenth year reenrollment randomized trial investigating the effects of childhood probiotics and calcium supplementation on height and weight at adolescence. Sci Rep. 2021 Jun 4;11(1):11860. doi: 10.1038/s41598-021-88819-y. PMID 34088920